CLINICAL TRIAL: NCT04250428
Title: Strategies to Increase Antenatal Iron and Folic Acid Supplementation and Malaria Prophylaxis in Rural South-central Côte d'Ivoire: Study Protocol of a Cluster Randomised Controlled Trial
Brief Title: Strategies to Increase Antenatal Iron and Folic Acid Supplementation and Malaria Prophylaxis
Acronym: AIFASMaP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Centre Suisse de Recherches Scientifiques en Cote d'Ivoire (Other)
Collaborators: Swiss Tropical & Public Health Institute (Other)
Responsible Party: Principal Investigator, Siaka Kone, Principal Investigator, Centre Suisse de Recherches Scientifiques en Cote d'Ivoire
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: TSS01021920
Record Dates: First submitted 2020-01-29; First posted 2020-01-31 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Antenatal Care
Keywords: antenatal iron and folic acid supplementation; malaria chemoprophylaxis; maternal and child health; Randomized controlled trial; Health and demographic surveillance site; Cost-effectiveness

STUDY DESIGN:
Intervention Model Description: This study is designed as a 3-arm parallel trial
Who Masked: Outcomes Assessor
Masking Description: Given the in-person nature pf both interventions, masking of subjects will not be possible. Interviewers conducting the final assessment will however be blinded to the treatment condition.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): Women in the control arm will have (standard) access to antenatal care.
- Demand intervention (Experimental): Women in this arm will receive a home visit by a study nurse at the beginning of their pregnancy that will inform them regarding the importance of iron and folic acid supplementation as well as malaria prophylaxis.
  Interventions: Behavioral: Demand intervention
- Supply intervention (Experimental): Women in this arm will get a monthly visit by study nurses. Women who did not obtain supplements or malaria prophyllaxis through routine antenatal care services will be directly provided with the supplements and malaria drugs by the study nurse.
  Interventions: Behavioral: Supply intervention

INTERVENTIONS:
Behavioral: Demand intervention — Women in the "demand intervention" arm will receive a home visit by a study nurse who will highlight the importance of supplementation and prophyllaxis to women. During this session, women will also be informed regarding side effects and the ideal timing of supplementation (after meals).
  Other Names: information intervention
  Arms: Demand intervention
Behavioral: Supply intervention — In order to directly test the importance of access barriers, we will deliver supplements as well as malaria chemo- prophyllaxis directly to women through home visits by study nurses.
  Other Names: Home delivery of supplements
  Arms: Supply intervention

SUMMARY:
Pregnancy increases the risk of malaria and nutritional deficiency. Despite some progress in ANC access over the past years, coverage of antenatal iron and folic acid supplementation (AIFAS) and intermittent preventive treatment of malaria in pregnancy (IPTp) remains low in many countries. The main objective of this research project is to identify the most effective ways to increase AIFAS and IPTp in low-income settings. We will assess the relative effectiveness of two strategies: the provision of information on the importance of AIFAS and IPTp for pregnant women (Intervention Arm I - demand side intervention), and the direct delivering of supplements and malaria drugs to women's homes (Intervention Arm 2 - supply side intervention). The two strategies will be tested through a small-randomized experiment with 720 pregnant women in the Taabo Health and Demographic Surveillance Site located in South-central Côte d'Ivoire. The primary outcome variable for the pilot study will be post-partum anemia and malaria infections. Secondary outcomes will be AIFAS and IPTp coverage as well as miscarriages, stillbirths and low birth weight deliveries as adverse birth outcomes.

DETAILED DESCRIPTION:
Background Despite major progress in antennal care (ANC) access over the past years, coverage of essential antenatal interventions remains limited in many low- and middle-income countries. At the same time, rates of maternal anemia and exposure to malaria in pregnancy remain high. In Côte d'Ivoire, 59% of pregnant women are estimated to be anemic (Hb< 110g/L), and only a minority of women receive antenatal iron supplementation consistently throughout their pregnancy and less than one third of women received intermittent preventive treatment of malaria in pregnancy (IPTp). Both interventions have been shown to be highly effective for reducing the risk of stillbirth, prematurity and low birth weight, and have been highlighted as essential for reducing the burden of malnutrition in the 2013 Lancet series. Low coverage rates of essential ANC interventions have been attributed to lacking demand from beneficiaries (e.g. low ANC attendance), weak early health system contact with women, limited funding, stock outages and ineffective management of supplies.

In general, limited coverage of essential health services as well as limited adherence to national protocol have been attributed to multiple challenges in the health system. These challenges include the lack of knowledge on importance of medication, interrupted supply and stock outs, high cost of care, lack of availability of services, and demand-side barriers such as distance, education, opportunity cost, and cultural and social barriers. To address these challenges successfully, a large number of community-based studies assessed a range of interventions including community-based distribution of drugs, vaccines, or other public health services. In 2018, a systematic review of strategies identified 28 studies evaluating the treatment coverage in community-based public health programs. These studies covered a range of different strategies, including community-based treatment, distributor incentives, distribution along kinship networks, intensified information, education, and communication activities, fixed-point delivery, conversion from school- to community-based delivery, and management by a non-governmental organization. Services delivered included community-based public child health programs such as vitamin A supplementation, child immunizations, and mass drug administration campaigns targeting neglected tropical diseases. The largest positive influence on treatment coverage was found for 4 strategies: community-directed distribution, incentives to increase distributor motivation, distribution along kinship networks and implementation of intensified IEC activities. A 2016 Cochrane review evaluated the effectiveness of community-based health education and household monetary incentives in child immunization coverage in low and middle-income countries (LMICs). Overall, health education at village meetings or at home, as well as household monetary incentives had only moderate-certainty evidence and little or no effect respectively on full immunization coverage. Vouchers have been widely used also to promote maternal and newborn health in low- and middle-income countries: a systematic review consolidated evidence from seven published systematic reviews on the effects of different types of cash transfers and vouchers on the use and quality of maternity care services. Positive findings were found, indicating that reproductive health voucher programs increased utilization of reproductive health services, improved quality of care, and improved population health outcomes. In another Cochrane review focusing directly on antenatal care, 34 randomized controlled trials testing community-based interventions to improve uptake of antenatal care (media campaigns, education or financial incentives for pregnant women), and health systems interventions (home visits for pregnant women or equipment for clinics) were identified. The review highlighted several potentially effective interventions, and suggested a combination of interventions for stronger impact.

Overall, evidence on the most effective ways to increase both IPTp and AIFAS remains mixed overall, with very few studies directly identifying cost-effective ways to increase coverage of both interventions. The objective of the proposed research is to assess both the cost, impact and relative cost-effectiveness of two of the most commonly used strategies in a rural low-income setting compared to the default system. This will help to identify the most effective ways to increase antenatal iron and folic acid supplementation (AIFAS) and IPT-p coverage among pregnant women in rural Cote d'Ivoire and similar settings.

Methods Study design The study will be designed as a cluster-randomized experiment with three arms: a control arm, an information or demand generation arm, and a direct distribution arm. The investigators expected to recruit approximately 240 pregnant women for each arm, for a total sample size of 720 women. This study will be carried out in the HDSS of Taabo in south-central Côte d'Ivoire. The Taabo HDSS has continuously monitored a population of approximately 45,000 since 2009. The pilot study will target 720 pregnant women across the 132 clusters constituting the HDSS monitoring area. The 132 clusters will be split into three groups: a control group (44 clusters), an information group (44 clusters), and a distribution of free supplements group (44 clusters).

Setting The proposed research will be implemented in the Taabo health and demographic surveillance site (HDSS), located some 160 km north-west of Abidjan, the economic capital of Côte d'Ivoire. The study area is mainly rural and covers a surface area of about 980 km2, but already displays clear signs of the epidemiological transition. The Taabo HDSS is situated in the health district of Tiassalé, which has an estimated population of 200,000 people. The HDSS area includes an urban setting (Taabo-Cité), 13 villages, and more than 100 small hamlets. Demographic data (i.e. pregnancy, birth, death, and in- and out-migration) are collected longitudinally at the individual and household level, usually in three data collection rounds per year. Deaths are reported by key informants and verbal autopsies are conducted using standard protocols to determine causes of death.

Main causes of death include malaria, HIV/AIDS, and tuberculosis. The HDSS population (approximately 45,000 individuals from 8,000 households) is predominantly Ivorian, with Akan as the main ethnic group. There are ten health facilities in the Taabo HDSS area: a 12-bed hospital in Taabo-Cité and nine health centers.

Selection of study participants Recruitment Pregnant women in the first trimester of their pregnancy, living in the HDSS with an age ≥15 and ≤ 49 years will be eligible to participate in this study. They should be registered as a member in the HDSS of Taabo and willing to provide one drop of blood for hemoglobin assessment and the rapid diagnostic malaria test. Key informants will be recruited by the study team in all areas to report pregnancies as early as possible to the study staff. Key informants will be given a reward of 1,000 CFA (USD 2) for each pregnancy reported. Once the study coordinator will be informed about a new pregnancy, he will then send out an interviewer to invite pregnant women to participate in the study. Conditional on women's consent, they will be enrolled in the study and a short baseline questionnaire will be conducted. Participants may decide not to continue participating in the study at any time for any reason if they wish to do so without any particular involvement. The investigator may decide to remove a participant from the study for reasons of ethical concerns or insufficient participant recruitment.

Participant Information and consent The investigators will use a separate informed consent form for this study. A general study participation consent form that will primarily cover the baseline and endline surveys, and consent forms for the two interventions. Mothers in the information (intervention) arm will be informed about the objective of this intervention. Mothers in the supplements arm will be informed about the objective of the arm as well as the package of this intervention. These intervention consent forms will be short and administered by study staff at the beginning of their first visit.

Pregnant women below 18 years old could be treated differently and depending on the situation. For non-emancipated mothers under 18, permission to participate in the study will be sought from a legal representative in the household. For illiterate mothers, the investigators will use a thumbprint instead of a signature on the consent form.

Intervention As part of this study, the investigators will conduct two interventions: a supply side intervention ("home delivery of iron and folic acid supplements and Sulfadoxine-pyrimethamine") and a demand side intervention ("providing information on the importance of IFAS and IPTp"). In the supply side intervention women will receive a monthly home visit by study staff. During this visit study staff will inform women about recommended ANC attendance and supplementation and inquire about supplements received. All women not having received supplements from their ANC visits will be provided with a monthly dose of iron and folic acid. Similarly, all women not having received SP will be directly provided SP together with additional information and instructions on how to take the medication. At the end of each visit, study staff will remind women about their next ANC appointment and remind them to take supplements daily. On the other hand, the demand side intervention focuses on empowering pregnant mothers to adopt appropriate health practices and health behavior. Health staff (midwives and nurses) will be trained to inform women on the importance of AIFAS as well as IPTp, and then visit all women in this arm at the beginning of their pregnancy. During this visit, the nurse will talk with participating women about the benefits, side-effects, and when, why, and how to take iron and folic acid supplements and SP. The nurse will also provide pregnant women with a phone number they can call in case they have questions related to ANC, supplements or IPTp.

Data collection

Data will be collected by a trained researcher team. In addition to the baseline collection, the investigators will collect detailed monitoring data on home visits as well as cost data for the two arms. To assess the relative effectiveness of each strategy, the investigators will conduct an endline survey within the first two weeks after delivery. The form to be used to conduct the endline survey among women will combine both information on prenatal supplementation and IPTp-SP (supplements, doses, period, frequency, and date, anemia and malaria status), socio-demographic characteristics (maternal age, education attainment, household assets), and pregnancy outcome (live birth, still birth, preterm birth, birth weight,). Given that the investigators expect women's self-report on AIFAS supplementation not be very accurate, the investigators will collect hemoglobin level and malaria infection rates as primary study outcome measures at endline. Hemoglobin levels will be assessed using HEMOCUE devices; malaria infection will be tested using standard Rapid Diagnostic Tests (RDTs). All endline surveys will be conducted by study nurses who are familiar with both test procedures.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women in the first trimester of their pregnancy, living in the HDSS with an age greater than or equal to 15 years.
* Be registered as a member in the HDSS of Taabo
* Willing to provide one drop of blood for hemoglobin assessment and the rapid diagnostic malaria test.
* Written informed consent
* Under 18 years with permission of legal representative

Exclusion Criteria:

* No written informed consent
* Under 18 years pregnant women without permission of legal representative
* Not registered as a member of the HDSS of Taabo

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 720 (Estimated)
Dates: Start 2020-02 (Estimated); Primary Completion 2021-05 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with a concentration of hemoglobin less than 11g/dL after delivery | Each mother will be enrolled in the study for approximately six months from the end of the first trimester to the endline survey conducted shortly after delivery. We will assess hemoglobin levels within the first two weeks after delivery
  Hemoglobin levels obtained assessed using HEMOCUE devices
Percentage of participants tested positive for malaria | Each mother will be enrolled in the study for approximately six months from the end of the first trimester to the endline survey conducted shortly after delivery. We will assess malaria infection within the first two weeks after delivery
  Malaria infection will be tested using standard Rapid Diagnostic Tests (RDTs).

REFERENCES:
- [Background] Christian P, Shrestha J, LeClerq SC, Khatry SK, Jiang T, Wagner T, Katz J, West KP Jr. Supplementation with micronutrients in addition to iron and folic acid does not further improve the hematologic status of pregnant women in rural Nepal. J Nutr. 2003 Nov;133(11):3492-8. doi: 10.1093/jn/133.11.3492. PMID 14608063
- [Background] Black RE, Victora CG, Walker SP, Bhutta ZA, Christian P, de Onis M, Ezzati M, Grantham-McGregor S, Katz J, Martorell R, Uauy R; Maternal and Child Nutrition Study Group. Maternal and child undernutrition and overweight in low-income and middle-income countries. Lancet. 2013 Aug 3;382(9890):427-451. doi: 10.1016/S0140-6736(13)60937-X. Epub 2013 Jun 6. PMID 23746772
- [Background] Bhutta ZA, Das JK, Rizvi A, Gaffey MF, Walker N, Horton S, Webb P, Lartey A, Black RE; Lancet Nutrition Interventions Review Group, the Maternal and Child Nutrition Study Group. Evidence-based interventions for improvement of maternal and child nutrition: what can be done and at what cost? Lancet. 2013 Aug 3;382(9890):452-477. doi: 10.1016/S0140-6736(13)60996-4. Epub 2013 Jun 6. PMID 23746776
- [Background] Sharma JB, Jain S, Mallika V, Singh T, Kumar A, Arora R, Murthy NS. A prospective, partially randomized study of pregnancy outcomes and hematologic responses to oral and intramuscular iron treatment in moderately anemic pregnant women. Am J Clin Nutr. 2004 Jan;79(1):116-22. doi: 10.1093/ajcn/79.1.116. PMID 14684407
- [Background] Trowbridge F, Martorell R. Summary and recommendations. J Nutr. 2002 Apr;132(4 Suppl):875S-9S. doi: 10.1093/jn/132.4.875S. PMID 11925502
- [Background] Brady J, Ho K, Kelley E, Clancy CM. AHRQs National Healthcare Quality and Disparities reports: an ever-expanding road map for improvement. Health Serv Res. 2007 Jun;42(3 Pt 1):xi-xxi. doi: 10.1111/j.1475-6773.2007.00736.x. No abstract available. PMID 17489895
- [Background] Ensor T, Cooper S. Overcoming barriers to health service access: influencing the demand side. Health Policy Plan. 2004 Mar;19(2):69-79. doi: 10.1093/heapol/czh009. PMID 14982885
- [Background] Ensor T, Dave-Sen P, Ali L, Hossain A, Begum SA, Moral H. Do essential service packages benefit the poor? Preliminary evidence from Bangladesh. Health Policy Plan. 2002 Sep;17(3):247-56. doi: 10.1093/heapol/17.3.247. PMID 12135990
- [Background] Deardorff KV, Rubin Means A, Asbjornsdottir KH, Walson J. Strategies to improve treatment coverage in community-based public health programs: A systematic review of the literature. PLoS Negl Trop Dis. 2018 Feb 8;12(2):e0006211. doi: 10.1371/journal.pntd.0006211. eCollection 2018 Feb. PMID 29420534
- [Background] Oyo-Ita A, Wiysonge CS, Oringanje C, Nwachukwu CE, Oduwole O, Meremikwu MM. Interventions for improving coverage of childhood immunisation in low- and middle-income countries. Cochrane Database Syst Rev. 2016 Jul 10;7(7):CD008145. doi: 10.1002/14651858.CD008145.pub3. PMID 27394698
- [Background] Bellows NM, Bellows BW, Warren C. Systematic Review: the use of vouchers for reproductive health services in developing countries: systematic review. Trop Med Int Health. 2011 Jan;16(1):84-96. doi: 10.1111/j.1365-3156.2010.02667.x. Epub 2010 Nov 2. PMID 21044235
- [Background] Mbuagbaw L, Medley N, Darzi AJ, Richardson M, Habiba Garga K, Ongolo-Zogo P. Health system and community level interventions for improving antenatal care coverage and health outcomes. Cochrane Database Syst Rev. 2015 Dec 1;2015(12):CD010994. doi: 10.1002/14651858.CD010994.pub2. PMID 26621223
- [Background] Kone S, Baikoro N, N'Guessan Y, Jaeger FN, Silue KD, Furst T, Hurlimann E, Ouattara M, Seka MC, N'Guessan NA, Esso EL, Zouzou F, Boti LI, Gonety PT, Adiossan LG, Dao D, Tschannen AB, von Stamm T, Bonfoh B, Tanner M, Utzinger J, N'Goran EK. Health & Demographic Surveillance System Profile: The Taabo Health and Demographic Surveillance System, Cote d'Ivoire. Int J Epidemiol. 2015 Feb;44(1):87-97. doi: 10.1093/ije/dyu221. Epub 2014 Nov 29. PMID 25433704
- [Background] Furst T, Silue KD, Ouattara M, N'Goran DN, Adiossan LG, N'Guessan Y, Zouzou F, Kone S, N'Goran EK, Utzinger J. Schistosomiasis, soil-transmitted helminthiasis, and sociodemographic factors influence quality of life of adults in Cote d'Ivoire. PLoS Negl Trop Dis. 2012;6(10):e1855. doi: 10.1371/journal.pntd.0001855. Epub 2012 Oct 4. PMID 23056662
- [Background] Kone S, Furst T, Jaeger FN, Esso EL, Baikoro N, Kouadio KA, Adiossan LG, Zouzou F, Boti LI, Tanner M, Utzinger J, Bonfoh B, Dao D, N'Goran EK. Causes of death in the Taabo health and demographic surveillance system, Cote d'Ivoire, from 2009 to 2011. Glob Health Action. 2015 May 8;8:27271. doi: 10.3402/gha.v8.27271. eCollection 2015. PMID 25959772
- [Derived] Kone S, Probst-Hensch N, Dao D, Utzinger J, Fink G. Improving coverage of antenatal iron and folic acid supplementation and malaria prophylaxis through targeted information and home deliveries in Cote d'Ivoire: a cluster randomised controlled trial. BMJ Glob Health. 2023 Apr;8(4):e010934. doi: 10.1136/bmjgh-2022-010934. PMID 37076197
- [Derived] Kone S, Utzinger J, Probst-Hensch N, Dao D, Fink G. Study protocol of a cluster randomized controlled trial of strategies to increase antenatal iron and folic acid supplementation and malaria prophylaxis in rural south-central Cote d'Ivoire. BMC Public Health. 2020 Oct 27;20(1):1609. doi: 10.1186/s12889-020-09626-0. PMID 33109138
- See also: World Malaria Report 2016 — http://apps.who.int/iris/bitstream/handle/10665/252038/9789241511711-eng.pdf?sequence=1
- See also: Enquête Démographique et de Santé et à Indicateurs Multiples de Côte d'Ivoire 2011-2012 — https://www.dhsprogram.com/pubs/pdf/FR272/FR272.pdf
- See also: Country Profile Indicators: Interpretation Guide — https://apps.who.int/iris/bitstream/handle/10665/44397/9789241599955_eng.pdf?ua=1